CLINICAL TRIAL: NCT00689429
Title: Natural History and Functional Outcome of Operatively Treated Open Pilon Fractures
Brief Title: Operatively Treated Open Pilon Fractures
Status: Completed | Type: Observational
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: DCG002; IRB# 27647EP
Record Dates: First submitted 2008-05-30; First posted 2008-06-03 (Estimated); Last update posted 2017-06-20 (Actual); Status verified 2017-06

CONDITIONS: Open Pilon Fractures
Keywords: Pilon Fractures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
A chart review will be performed to extrapolate information including sex, height, weight, date/time admitted to HMC, injury data, comorbidities, fracture pattern, antibiotic usage, surgical history, wound history, fracture healing, and length of time to return to work. Dr.'s Goodspeed and Reid will conduct a radiographic review independently for each subject, classifying all fractures according to the Orthopaedic Trauma Association classification guide. If a discrepancy in classification is found, then both will discuss together and come to a consensus.

DETAILED DESCRIPTION:
After patients are identified with the Orthopaedic Surgical Database, letters will be sent to those patients who meet inclusion/exclusion criteria informing them of the study and that they will be contacted by the research associate in 1-2 weeks. The research associate will telephone the patient to discuss the study and answer any questions they may have. Dr. Goodspeed will also be available to answer any questions. The research associate with obtain verbal consent and proceed by asking questions from the Short Musculoskeletal Function Assessment Injury and Arthritis Survey, and the Foot and Ankle Outcomes Questionnaire. The medical student will then perform a chart review to extrapolate information including sex, height, weight, date/time admitted to HMC, injury data, comorbidities, fracture pattern, antibiotic usage, surgical history, wound history, fracture healing, and length of time to return to work. Dr.'s Goodspeed and Reid will conduct a radiographic review independently for each subject, classifying all fractures according to the Orthopaedic Trauma Association classification guide. If a discrepancy in classification is found, then both will discuss together and come to a consensus.

Functional outcomes data will be measured by the Short Musculoskeletal Function Assessment Injury and Arthritis Survey and the Foot and Ankle Outcomes Questionnaire. Radiographic Classifications will be determined according to the Orthopaedic Trauma Association's classification guide.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to the Hershey Medical Center with a primary diagnosis of an open pilon fracture and surgically treated between 1/1/2000 and 12/31/2007.
* Temporization of the fracture may be performed elsewhere or by other orthopaedists at the Hershey Medical Center. Definitive surgery must be performed by Dr.'s David Goodspeed, J. Spence Reid, or Robert Simpson.

Exclusion Criteria:

* closed pilon fracture or pathological fracture; definitive fracture fixation performed outside the Hershey Medical center or by a surgeon other than Dr.'s David Goodspeed, J. Spence Reid, and Robert Simpson; patient is diagnosed with active infection at the time of first surgery at the Penn State Hershey Medical Center; patient is less than 18 years of age at the time of definitive surgery;
* patient is mentally compromised and unable to give consent;
* does not cooperate with survey data acquisition; patient is deceased;
* patient presented with significant ipsilateral leg fracture or injury at anytime within the time frame of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (18 years and older) patients treated with definitive open reduction and fixation of open pilon fractures between 2000 - 2007 at Hershey Medical Center.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2008-05; Primary Completion 2010-04-09 (Actual); Study Completion 2010-04-09 (Actual)

PRIMARY OUTCOMES:
Functional outcomes data will be measured by the Short Musculoskeletal Function Assessment Injury and Arthritis Survey and the Foot and Ankle Outcomes Questionnaire. Radiographic Classifications will be determined. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: David C Goodspeed, MD, Principal Investigator — Penn State Hershey Medical Center and College of Medicine
Locations (1):
- Penn State Hershey Medical Center and College of Medicine, Hershey, Pennsylvania, United States